CLINICAL TRIAL: NCT06198088
Title: Effects of Proprioception Neuromuscular Facilitation Technique in Children With Post Fracture Elbow Stiffness
Brief Title: Effects of PNF Technique in Children With Post Fracture Elbow Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0744
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The patient in the experiment group will PNF techniques (hold relax) the participants who were assigned for post traumatic stiffness of the elbow with baseline treatment (heating pad), stretching applied for 30 sec then relaxation time 10 sec, 5 repetition were given in a session for 5 days a week for 4 weeks.
  Interventions: Other: PNF techniques
- control group (Other): exercise therapy range of motion, stretching and strengthening were applied with heating pad as baseline treatment. 5 repetition were given in a session for 5 days a week for 4 week.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: PNF techniques — The patient in the experiment group will PNF techniques (hold relax) the participants who were assigned for post traumatic stiffness of the elbow with baseline treatment (heating pad), stretching applied for 30 sec then relaxation time 10 sec, 5 repetition were given in a session for 5 days a week for 4 weeks.
  Arms: experimental group
Other: Exercise therapy — exercise therapy range of motion, stretching and strengthening were applied with heating pad as baseline treatment. 5 repetition were given in a session for 5 days a week for 4 week.
  Arms: control group

SUMMARY:
Daily living activities are an essential part of a child's development, providing endless opportunities for play, learning, and imaginative expression. The desired result as the child get bored after a while so we use it for benefits. Proprioceptive Neuromuscular Facilitation is a stretching technique utilized to improve muscle elasticity and has been shown to have a positive effect on active and passive range of motions. In clinical settings, PNF is already utilized by therapists to restore functional range of motion (ROM) and increase strength in patients who have sustained soft tissue damage or received invasive surgeries.

DETAILED DESCRIPTION:
This Randomized clinical trial study will be conducted in THQ hospital Arifwala/DHQ pakpattan with calculated sample size 26. Study will be approved by ethical committee. After that informed consent will be taken and patients will be randomly assigned to (Group A) control group these individuals will receive Maitland's mobilization with everyday object activities (Group B) experimental group (these individuals will receive baseline treatment and PNF technique ) frequency will be 5 session per week of 30 min and duration is of 4 weeks. Ranges will be assessed by Goniometry DASH outcome measure scale will use to assess functional activity. Data will be analyzed by SPSS latest version.

ELIGIBILITY:
Inclusion Criteria:

* Children Age 3-7 years
* Either gender
* Contracture 4-8 weeks post traumatic injuries.
* Post-operative

Exclusion Criteria:

* Burn contracture
* Contracture due to neurological conditions
* Dupytren's contracture, Volkmann's contracture etc.
* Contracture more than 8 week

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
DASH | 4 weeks
  DASH is a 30-item self-report questionnaire designed to assess musculoskeletal disorders of upper limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Sumaira Bibi, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sim G, Fleming J, Glasgow C. Mobilizing orthoses in the management of post-traumatic elbow contractures: A survey of Australian hand therapy practice. J Hand Ther. 2021 Jan-Mar;34(1):90-99. doi: 10.1016/j.jht.2019.12.014. Epub 2020 Mar 7. PMID 32156579
- See also: Mobilizing orthoses in the management of post-traumatic elbow contractures — https://pubmed.ncbi.nlm.nih.gov/32156579/.